CLINICAL TRIAL: NCT02258308
Title: Medicaid Asthma Home Visit Project: Improving Health and Reducing Costs of Health Care for Children With Asthma
Brief Title: CDC Medicaid Asthma Home Visit Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health - Seattle and King County (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHSKC
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHW intervention (Experimental): The CHW intervention is in-home education and support by a community health worker (CHW). At the first home visit, the CHW assesses the participant's knowledge and skills related to asthma self-management, current status of the child's asthma, and resources and support for asthma self-management using a baseline questionnaire. The CHW will inspect the home environment using an Environmental Home Checklist to identify environmental triggers that can cause asthma symptoms and affect asthma control. The CHW makes up to three follow-up visits and two telephone visits during the year the participant is in the study. Participants receive resources to help them control asthma: vacuum cleaner, dust covers for a pillow and mattress and a "green" cleaning kit with cleaning supplies.
  Interventions: Behavioral: CHW intervention
- control (No Intervention): The control group receives standard asthma care, as provided by a primary health care provider. When the intervention period is over, the control group receives one visit with a CHW and the resources provided to the intervention group participants.

INTERVENTIONS:
Behavioral: CHW intervention — Home education and support for asthma self management
  Arms: CHW intervention

SUMMARY:
Asthmatic children age 3-17 from low income households in King County are randomly assigned into a community health worker (CHW) intervention group and a control group. The intervention is in-home education and support related to asthma self-management. The main outcome measures are asthma symptom-free days, caretaker's asthma-related quality of life score, and health care utilization for asthma measured at baseline and 12 months after baseline enrollment.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Potentially eligible subjects come from lists generated by health plans (Community Health Plan of Washington and Molina, who insure the majority of Medicaid enrollees in King County), individuals referred by primary care providers, and self referral. Eligible subjects that agree to participate are randomly assigned into a CHW intervention group or a control group. We expected to complete the study with 200 in each group.

The intervention is in-home education and support by a community health worker (CHW). At the first home visit, the CHW assesses the participant's knowledge and skills related to asthma self-management, current status of the child's asthma, and resources and support for asthma self-management using a baseline questionnaire. The CHW inspects the home environment using an Environmental Home Checklist to identify environmental triggers that can cause asthma symptoms and affect asthma control. The CHW makes up to three follow-up visits and two telephone visits during the year the participant is in the study. Participants receive resources to help them control asthma, including vacuum cleaner, dust covers for a pillow and mattress and a "green" cleaning kit with cleaning supplies.

The control group receives standard asthma care, as provided by a primary health care provider during the 12 months after enrollment. When the intervention period is over, the control group receives one visit with a CHW and the resources provided to the intervention group participants.

The main outcome variables include asthma symptom-free days, caretaker asthma-related quality of life, and urgent health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* caretaker is age 18 or older and child is age 3-17
* have not controlled as thma
* residence in King County
* spoken language is English or Spanish
* Child is enrolled in a Medicaid managed care health plan offered by Community Health Plan of Washington (CHPW) or Molina Health Plan of Washington, Inc (Molina).

Exclusion Criteria:

* Parent/guardian plans to move out of King County within the next year or lacks permanent housing.
* Parent/guardian has a mental or physical disability making it impossible to participate in the protocols.
* The household appears to be unsafe for visitation by the CHW.
* The child has other serious chronic medical conditions (e.g. poorly controlled sickle cell disease, cystic fibrosis) that cause sufficient limitation in functional status so that that asthma control is not a priority.
* The family is enrolled in another asthma research study within the past three years. This is to avoid the potential confounding effect from other studies.
* The child is in foster care or group care settings.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Asthma symptom free days | last 14 days
  14 - During the past 14 days (that is, during the past fourteen 24 hour periods that include daytime and nighttime), on how many DAYS did your child have any asthma symptoms, such as wheezing, coughing, tightness in the chest, shortness of breath, waking up at night because of asthma symptoms, or slowing down of usual activities because of asthma?
Caretaker quality of life | last week
  Juniper Mini Asthma Quality of Life Questionnaire
Health care utilization for asthma | 12 months
  number of unscheduled clinic visits+emergency department visits+hospitalization for asthma
cost analysis | 12 months
  costs associated with health care utilization for asthma

SECONDARY OUTCOMES:
nights with asthma symptoms | 14 days
  During the nighttime in the past 14 nights, how many nights did your child wake up because of asthma symptoms such as wheezing, shortness of breath, or tightness in the chest, or cough?
days with activity limitation due to asthma | 14 days
  During the past 14 days, how many days did your child have to slow down or stop his/her play or usual activities or missed school because of asthma, wheezing or tightness in the chest, or cough.
days used asthma rescue medicine | 14 days
  During the past 14 days, about how many days did your child use asthma rescue medicine (sometimes called a quick relief medicine) such as albuterol, proventil, or ventolin?
asthma episodes | 3 months
  During the past three months, about how many asthma episodes did your child have?
asthma control level | 14 days
  (% with well controlled asthma and % with very poorly controlled asthma)

REFERENCES:
- [Result] Campbell JD, Brooks M, Hosokawa P, Robinson J, Song L, Krieger J. Community Health Worker Home Visits for Medicaid-Enrolled Children With Asthma: Effects on Asthma Outcomes and Costs. Am J Public Health. 2015 Nov;105(11):2366-72. doi: 10.2105/AJPH.2015.302685. Epub 2015 Aug 13. PMID 26270287